CLINICAL TRIAL: NCT02520180
Title: A Prospective Multicenter Post Market Trial to Assess the Safety and Effectiveness of the Firehawk™ Rapamycin Target Eluting Cobalt Chromium Coronary Stent System (Firehawk™ Stent System) for the Treatment of Atherosclerotic Lesion(s)
Brief Title: Non-inferiority Study Comparing Firehawk Stent With Abbott Xience Family Stent (TARGET-AC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TARGET AC
Record Dates: First submitted 2015-07-29; First posted 2015-08-11 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Firehawk™ stent system (Experimental): MicroPort Firehawk™ stent system
  Interventions: Device: Firehawk™ stent system
- Xience family Everolimus-Eluting Stent (Active Comparator): Abbott Xience family Everolimus-Eluting Stent
  Interventions: Device: Abbott Xience family Everolimus-Eluting Stent

INTERVENTIONS:
Device: Firehawk™ stent system — MicroPort Firehawk™ biodegradable polymer rapamycin target eluting stent
  Other Names: MicroPort Firehawk™ rapamycin target eluting stent
  Arms: Firehawk™ stent system
Device: Abbott Xience family Everolimus-Eluting Stent — Abbott Xience family Everolimus-Eluting Stent
  Arms: Xience family Everolimus-Eluting Stent

SUMMARY:
Purpose The TARGET All comers trial is a prospective, multicenter, randomized, two-arm, non-inferiority, open-label study with 1656 patients at 20 centers in Europe. The study is a "real world, all comers" study.

DETAILED DESCRIPTION:
Primary objective: to compare the MicroPort Medical (Group) Co., Ltd Firehawk™cobalt chromium coronary stent ( rapamycin target eluting ) system with abluminal grooves containing a biodegradable polymer with the Abbott XIENCE family EES (Everolimus-Eluting stent) system with respect to cardiac death, myocardial infarction (not clearly attributable to a non-target vessel), Target Lesion Revascularization at 1 year in a "real world" patient population.

ELIGIBILITY:
Inclusion Criteria:

* Minimal age 18 years
* Symptomatic coronary artery disease
* Patient acceptable candidate for treatment with drug eluting stent in accordance with applicable guidelines
* Presence of one or more coronary artery stenosis >50% with reference diameter 2.25-4.0mm which can be covered by one or multiple stents
* Patient indication, lesion length and vessel diameter according to 'Instructions for Use' of study stents
* Patient is willing and able to cooperate with study procedures and required follow up visits and patient or legal representative has been informed and agrees by signing EC approved written informed consent

Exclusion Criteria:

* Women of childbearing potential who do not have a negative pregnancy test within 7 days before procedure and women who are lactating
* Known intolerance to aspirin, clopidogrel or ticlopidin, heparin, cobalt, nickel, chromium, molybdenum, polymer coatings, Sirolimus, Everolimus, or contrast material
* Participating in other trial before reaching primary endpoint
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1653 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure | 12 months
  Percentage of participants that had either Cardiac Death, Myocardial Infarction (not clearly attributable to a non-target vessel)or Target Lesion Revascularization (TLR, clinically indicated) after one year

SECONDARY OUTCOMES:
In-stent late loss | 13 months
  In-stent late loss at 13 months post-procedure as measured by quantitative coronary angiography (QCA)
stent struth Neointimal thickness | 3 months
  stent struth Neointimal thickness at 3 months measured by Optical Coherence Tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: William Wijns, MD, PhD, Study Chair — VZW Cardiovascular Research Center Aalst; Andreas Baumbach, MD, Principal Investigator — Bristol Heart Institute/University Hospitals Bristol NHS Foundation Trust,UK; Alexandra Lansky, MD, Principal Investigator — Yale Cardiovascular Research Group,USA
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu B, Saito Y, Baumbach A, Kelbaek H, van Royen N, Zheng M, Morel MA, Knaapen P, Slagboom T, Johnson TW, Vlachojannis G, Arkenbout KE, Holmvang L, Janssens L, Ochala A, Brugaletta S, Naber CK, Anderson R, Rittger H, Berti S, Barbato E, Toth GG, Maillard L, Valina C, Buszman P, Thiele H, Schachinger V, Lansky A, Wijns W; TARGET AC Investigators. 2-Year Clinical Outcomes of an Abluminal Groove-Filled Biodegradable-Polymer Sirolimus-Eluting Stent Compared With a Durable-Polymer Everolimus-Eluting Stent. JACC Cardiovasc Interv. 2019 Sep 9;12(17):1679-1687. doi: 10.1016/j.jcin.2019.05.001. Epub 2019 May 22. PMID 31129092
- [Derived] Lansky A, Wijns W, Xu B, Kelbaek H, van Royen N, Zheng M, Morel MA, Knaapen P, Slagboom T, Johnson TW, Vlachojannis G, Arkenbout KE, Holmvang L, Janssens L, Ochala A, Brugaletta S, Naber CK, Anderson R, Rittger H, Berti S, Barbato E, Toth GG, Maillard L, Valina C, Buszman P, Thiele H, Schachinger V, Baumbach A; TARGET All Comers Investigators. Targeted therapy with a localised abluminal groove, low-dose sirolimus-eluting, biodegradable polymer coronary stent (TARGET All Comers): a multicentre, open-label, randomised non-inferiority trial. Lancet. 2018 Sep 29;392(10153):1117-1126. doi: 10.1016/S0140-6736(18)31649-0. Epub 2018 Sep 3. PMID 30190206